CLINICAL TRIAL: NCT01867320
Title: Pilot Study of Raltegravir, an Integrase Inhibitor, in Human T-Cell Lymphotrophic Virus-1(HTLV-1) Associated Myelopathy, Tropical Spastic Paraparesis (HAM/TSP)
Brief Title: Raltegravir for HAM/TSP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130135; 13-N-0135
Record Dates: First submitted 2013-05-21; First posted 2013-06-04 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: HTLV-I Infection
Keywords: PVL; Immune; Activation; HTLV-1; HTLV-1 Associated Myelopathy
MeSH Terms: conditions — HTLV-I Infections; Paraparesis, Tropical Spastic | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raltegravir (Experimental): Raltegravir at 400mg by mouth twice daily in an initial 6 months treatment phase, followed by an additional 9 months post treatment phase.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir at 400mg by mouth twice daily in an initial 6 months treatment phase, followed by an additional 9 months post treatment phase.

SUMMARY:
Background:

- Human T-cell lymphotropic virus type 1 associated myelopathy/tropical spastic paraparesis (HAM/TSP) is an infection of the spinal cord. The infection is caused by a virus that has been known to cause cancers like leukemia and lymphoma. It causes a weakening of the legs. Researchers want to see if raltegravir, a drug for treating human immunodeficiency virus (HIV), can be used to treat HAM/TSP. They will see if the drug can reduce the amount of virus in the blood of people with HAM/TSP.

Objectives:

- To see if raltegravir can reduce the viral load of people with HAM/TSP.

Eligibility:

- Individuals at least 18 years of age who have HAM/TSP.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected. Imaging studies will be performed. A lumbar puncture will also be taken.
* Participants will take the study drug twice a day for 6 months. They will note each dose in a study diary, as well as any side effects.
* At the 6-month visit, participants will stop taking the study drug. They will have a physical exam and blood samples, as well as other tests.
* Participants will have two further exams 9 months and 15 months after starting the study drug. They will have a physical exam and blood samples, as well as other tests.

DETAILED DESCRIPTION:
Objective:

In this pilot study, we wish to determine the effects of Raltegravir, a clinically approved HIV-1 integrase inhibitor, on HTLV-1 proviral load (PVL) in patients with HTLV-1 associated myelopathy / tropical spastic paraparesis (HAM/TSP). We will also provide safety and tolerability information on Raltegravir use in this condition and examine the correlation of immune activation markers in HAM/TSP with the effects of Raltegravir on the PVL.

Study population:

HAM/TSP, a relentlessly progressive and disabling myelopathy, occurs in up to 3% of HTLV-1 infected subjects. It results from immune-mediated bystander damage of the neural tissues in association with an elevated PVL. In fact, a high PVL is considered to be the main risk factor for developing HAM/TSP as the risk of disease rises exponentially once the PVL exceeds 1 %. Currently there is no effective treatment for HAM/TSP.

There is evidence that active HTLV-1 replication, through the retroviral life cycle with new virus integration, is occurring in vivo and contributes to the total HTLV-1 PVL in infected subjects. Recently it was shown that Raltegravir could inhibit cell-free and cell-to-cell transmission of HTLV-1 in vitro. Given the substantial clinical experience with its use in HIV-1 infection and particularly its excellent safety profile, this agent is an attractive therapeutic option for patients with HAM/TSP, either alone or in combination with immunomodulatory treatment. In this pilot study we wish to determine the effects of Raltegravir in vivo on HTLV-1 PVL and immune activation markers in patients with HAM/TSP.

Design:

In this 15 months single center, single arm, open label, baseline versus treatment pilot clinical trial, sixteen subjects with HAM/TSP will receive Raltegravir at 400mg by mouth twice daily in an initial 6 months treatment phase, followed by an additional 9 months post treatment phase. Outcome measures will be collected every 3 months for the duration of the study.

Outcome measures:

The primary outcome measure is HTLV-1 proviral load, which will be measured by quantitative PCR. Secondary outcome measures include safety and tolerability of Raltegravir, which will be assessed by clinical exam and standardized neurological disability scales as well as clinical laboratory studies. In addition, viral and immunologic outcome measures investigating the impact of Raltegravir on HTLV-1 biology and its effects on immune function will be measured including HTLV-1 proviral load in different lymphocyte populations, the number of long terminal repeat (LTR) circles and HTLV-1 mRNA expression levels in freshly isolated PBMC, assays of spontaneous lymphoproliferation and T-cell phenotype analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 years or older
* Diagnosis of HAM/TSP as defined by WHO criteria, including a positive HTLV-1 EIA and confirmatory Western Blot.
* Patient must be willing and able to comply with all the aspects of trial design and follow-up.
* Patients must be able to provide informed consent
* If able to become pregnant or to father a child, agreeing to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation, or vasectomy) for the duration of treatment arm of the study

EXCLUSION CRITERIA:

* Alternative diagnoses that can explain neurological disability
* Clinically significant medical disorders that, in the judgment of the investigators might expose the patient to undue risk of harm confound study outcomes or prevent the patient from completing the study. Examples of such conditions include but are not limited to poorly controlled cardiopulmonary conditions such as congestive heart failure, asthma or uncontrolled hypertension.
* Patient has received immunomodulatory/immunosuppressive therapy (including steroids) in the preceding 6 months.
* Patient with known myopathy or risk factors for CK elevation including being on other drugs known to cause myopathy or rhabdomyolysis.
* Pregnant or lactating women.
* Patient has received other investigational drugs within 6 months before enrollment
* Positive serological evidence of HIV, HTLV-II, Hepatitis B or C.
* Abnormal screening/baseline blood tests exceeding any of the limits defined below:

  * Serum alanine transaminase (ALT) or aspartate transaminase (AST) levels greater than 3 times the upper limit of normal values; total bilirubin > 2.0mg/dl; Serum amylase or lipase levels greater than twice the upper limit of normal values; serum creatine phosphokinase (CK) level exceeding 3 xULN and confirmed on repeat testing in 2 weeks.
  * Platelet count < 75,000/mm(3)
  * Serum creatinine level > 2.0 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
HTLV-1 Proviral load, which will be measured by quantitative PCR | month 6 compared to pretreatment value
  The primary outcome measure is HTLV-1 proviral load in the peripheral blood mononuclear cells (PBMCs) measured by Taqman at month 6 compared to pretreatment value.

SECONDARY OUTCOMES:
Safety and tolerability of Raltegravir | each patient visit
  Safety and tolerability will be assessed at each patient visit by full interim history, physical exam and clinical bloodwork. Neurologic safety will be specifically assessed by Standardized neurologic examination and scoring relevant to HAM/TSP

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jacobson, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Araujo AQ, Andrade-Filho AS, Castro-Costa CM, Menna-Barreto M, Almeida SM. HTLV-I-associated myelopathy/tropical spastic paraparesis in Brazil: a nationwide survey. HAM/TSP Brazilian Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Dec 15;19(5):536-41. doi: 10.1097/00042560-199812150-00014. PMID 9859969
- [Background] Asquith B, Hanon E, Taylor GP, Bangham CR. Is human T-cell lymphotropic virus type I really silent? Philos Trans R Soc Lond B Biol Sci. 2000 Aug 29;355(1400):1013-9. doi: 10.1098/rstb.2000.0638. PMID 11186302
- [Background] Aye MM, Matsuoka E, Moritoyo T, Umehara F, Suehara M, Hokezu Y, Yamanaka H, Isashiki Y, Osame M, Izumo S. Histopathological analysis of four autopsy cases of HTLV-I-associated myelopathy/tropical spastic paraparesis: inflammatory changes occur simultaneously in the entire central nervous system. Acta Neuropathol. 2000 Sep;100(3):245-52. doi: 10.1007/s004019900170. PMID 10965793
- [Derived] Enose-Akahata Y, Billioux BJ, Azodi S, Dwyer J, Vellucci A, Ngouth N, Nozuma S, Massoud R, Cortese I, Ohayon J, Jacobson S. Clinical trial of raltegravir, an integrase inhibitor, in HAM/TSP. Ann Clin Transl Neurol. 2021 Oct;8(10):1970-1985. doi: 10.1002/acn3.51437. Epub 2021 Sep 25. PMID 34562313
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-N-0135.html